CLINICAL TRIAL: NCT02550743
Title: BrUOG 302:BYL719, Capecitabine and Radiation for Rectal Cancer: A Brown University Oncology Research Group Phase I Study
Brief Title: BrUOG 302:BYL719, Capecitabine and Radiation for Rectal Cancer: A Brown University Oncology Research Group Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accural
Sponsor: howard safran (Other)
Collaborators: Brown University (Other); Lifespan (Other); Novartis Pharmaceuticals Corporation (Financial supporter) (Unknown)
Responsible Party: Sponsor-Investigator, howard safran, Principal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 302
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Rectal Cancer
Keywords: Stage II; Stage III; Stage IV; metastatic
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis | interventions — Alpelisib; Capecitabine; Radiation

STUDY DESIGN:
Intervention Model Description: This is a phase I dose escalation study adding BYL719 to standard capecitabine and radiation.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose 1 (Experimental): BYL719, capectabine and radiation Dose BYL719: 200mg/day
  Interventions: Drug: BYL719; Drug: Capecitabine; Radiation: Radiation
- Dose 2 (Experimental): BYL719, capectabine and radiation Dose BYL719: 250mg/day
  Interventions: Drug: BYL719; Drug: Capecitabine; Radiation: Radiation
- Dose 3 (Experimental): BYL719, capectabine and radiation Dose BYL719: 300mg/day
  Interventions: Drug: BYL719; Drug: Capecitabine; Radiation: Radiation
- Dose -1 (Experimental): BYL719, capectabine and radiation Dose BYL719: 150mg/day
  Interventions: Drug: BYL719; Drug: Capecitabine; Radiation: Radiation

INTERVENTIONS:
Drug: BYL719
Drug: Capecitabine
  Other Names: Xeloda
Radiation: Radiation

SUMMARY:
The primary goal of this Brown University Oncology Research Group is to determine that a safe dose of BYL719 can be administered with capecitabine and radiation in patients with rectal cancer. Therefore, the threshold of success for this phase I study is to establish safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven adenocarcinoma of the rectum with no evidence of distant metastases.
* The tumor must be clinically Stage II (T3-4 N0) or stage III (N+). Stage of the tumor may be determined by CT scan, endorectal ultrasound or MRI. (For patients receiving chemotherapy prior to protocol chemoradiation, the initial clinical stage applies. CT/MRI/PET should be performed within 2 months of study entry to exclude disease progression.). For the MTD expansion phase only: patients who are stage IV, and in whom it is planned to administer capecitabine and radiation then have a resection of their rectal cancer, are also eligible.
* Measurable disease not required at baseline. Patient's without measurable disease may be enrolled as long as they clinically meet stage II or III criteria or for MTD expansion phase: also stage IV.
* Patients must not have received pelvic radiation for rectal cancer, or prior pelvic radiation for any other malignancy that would prevent the patient from receiving the required radiation treatments for this study. (Patients may receive neoadjuvant chemotherapy prior to study chemoradiation)
* Patients must not have an active concurrent invasive malignancy. Patients with prior malignancies, including invasive colon cancer, are eligible if they are deemed by their physician to be at low risk for recurrence. For example, patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 3 years prior to registration.
* Patients must be > 18 years of age,
* ECOG performance status 0-1
* Neutrophil Count >1,000/µl, platelets >100,000/µl, total bilirubin < 1.5 x< ULN ULN (except for patients with Gilbert's syndrome who may only be included if total bilirubin is < 3xULN with direct bilirubin within normal range), ALT <2.5xULN, AST < 2.5xULN, creatinine <1.5xULN, fasting plasma glucose < 140 mg/dL and HbA1c < 6.4% (both criteria have to be met), anemia > 9.0g/dL.Potassium, Calcium and Magnesium (corrected for albumin) within normal range or < grade 1 if determined not clinically significant by treating investigator. INR < 1.5
* Patient is able to swallow and retain oral medication.
* Left ventricular ejection fraction within normal >50%
* Signed informed consent and is able to comply with study and/or follow- up procedures.
* QTcF <480 msec
* Patients history of diarrhea has been review and patient has been informed of potential study drug induced diarrhea and management. This must be documented by treating MD. See section 5 for baseline assessments of patient history of diarrhea.

Exclusion Criteria:

* Patient has a known hypersensitivity to any of the excipients of BYL719 (alpelisib)
* Suspected or confirmed metastatic disease including CNS involvement. For stage IV patients: CNS involvement.
* Patient with clinically manifest diabetes mellitus, or documented steroid induced diabetes mellitus
* Patient with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with colostomies are allowed unless colostomy is for one of the precluded reason above.
* Patient who has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient who has had systemic therapy within 4 weeks of starting study treatment (6 weeks for nitrosoureas or mitomycin C)
* Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or in the investigators opinion who has not recovered from side effects of such procedure
* Patient has any of the following cardiac abnormalities: A. symptomatic Congestive heart failure i. history of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy ii. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) B. myocardial infarction < 6 months prior to enrollment C. unstable angina pectoris D. serious uncontrolled cardiac arrhythmia E. symptomatic pericarditis F. QTcF > 480 msec on the screening ECG (using the QTcF formula)
* Patient who is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment. To be documented and submitted to BrUOG with registration. Please refer to appendices F and G.
* Patient who has participated in a prior investigational cancer treatment study within 30 days prior to enrollment. This refers to treatment not follow-up.
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed. To be documented and submitted to BrUOG with registration. Eliquis is allowed.
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment. Switching to a different medication prior to registration is allowed; (Refer to Section Concomitant Medication, Appendix F and G).
* Patient with known positive serology for human immunodeficiency virus (HIV)
* Patient with any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow oral medication, social/psychological complications, chronic active hepatitis, severe hepatic impairment etc
* Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgment, contraindicate patient participation in the individual patient program (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL). Pregnancy test not required for patients who are considered post-menopausal and not of childbearing potential as defined below.

Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

For women with therapy-induced amenorrhea, oophorectomy or serial measurements of FSH and/or estradiol are needed to ensure postmenopausal status.

* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

  1. Sexually active males (unless surgically sterilized at least 6 months prior to screening) should use a condom during intercourse while taking drug and for 6 months after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. The use of spermicidal foam is also highly suggested to be used with a condom as another form of protection. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. Males should be cautioned to not donate sperm while actively receiving treatment on study.
  2. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through 6 months after the final dose of study treatment.
* Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, Medical Marijuana and ginseng. Patients need to stop using these herbal medications 7 days prior to first dose of study drug.
* Patient must not eat or drink Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pummelos, starfruits and cranberry juice from 7 days prior to the first dose of study drug and during the entire study treatment
* Patient is currently receiving or has received systemic corticosteroids < 2 weeks prior to day 1 of study drug, or who has not fully recovered from side effects of treatment. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Patient is concurrently using other anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (1):
- Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1: BYL719, capectabine and radiation Dose: 200mg/day
  BYL719
  Capecitabine
  Radiation
- Dose 2: BYL719, capectabine and radiation Dose: 250mg/day
  BYL719
  Capecitabine
  Radiation
- Dose 3: BYL719, capectabine and radiation Dose: 300mg/day
  BYL719
  Capecitabine
  Radiation
- Dose -1: BYL719, capectabine and radiation Dose: 150mg/day
  BYL719
  Capecitabine
  Radiation
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose -1
Started | 3 | 3 | 1 | 0
Completed | 3 | 3 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no patients were registered to dose level -1
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose -1 | Total
Number analyzed (Participants) | 3 | 3 | 1 | 0 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 1 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [36 to 48] | 50 [40 to 58] | 54 [54 to 54] |  | 47.6 [36 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 3
  Male | 2 | 2 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 0 | 0 | 6
  Unkown | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of BYL719
Time Frame: approximately 6 weeks
Measure: Number; unit: mg
Groups:
- Maximum Tolerated Dose of BYL719: BYL719, capectabine and radiation
Arm/Group | Maximum Tolerated Dose of BYL719
Number analyzed (Participants) | 7
mg | NA — insufficient number of participants with events to determine MTD

2. Secondary Outcome: Pathologic Complete Response for Patients With Rectal Cancer
Description: Pathologic complete response is defined as the lack of all signs of cancer in tissue samples removed during surgery or biopsy after treatment with radiation or chemotherapy.
Time Frame: Approximately 6-10 weeks post treatment
Population: No patients enrolled on dose -1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose -1
Number analyzed (Participants) | 3 | 3 | 1 | 0
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent through 30-days post treatment, an average of 3 months
Description: No patients were enrolled to dose -1.
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose -1
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=3) | Dose 2 (N=3) | Dose 3 (N=1) | Dose -1 (N=0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=3) | Dose 2 (N=3) | Dose 3 (N=1) | Dose -1 (N=0)
anemia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
dehydration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
erythema multiforme (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FPG-hyperglycemia (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HTN (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
pain abdominal (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
pain rectal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
pain vaginal (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Radiation (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
peripheral sensory neuropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALT (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vomit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypermagnesium (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pain perineal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders other: rectal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
infection (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pelvic pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT02550743/Prot_SAP_ICF_000.pdf